CLINICAL TRIAL: NCT04574180
Title: Can Zirconia Crown be the First Restorative Choice After Endodontic Treatment for Primary Teeth?
Brief Title: Can Zirconia Crown be the First Choice for Primary Teeth?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Aslı GÜÇLÜ, Assocciate Prof, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSA-2017-6723
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dental Caries in Children
Keywords: zirconia; crown; endodontic; pediatric
MeSH Terms: interventions — Crowns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Zirconia crown anterior (NuSmile, Houston, Texas, USA).
  Interventions: Other: Dental Crown
- Group 2 (Active Comparator): Zirconia crown posterior (NuSmile, Houston, Texas, USA).
  Interventions: Other: Dental Crown
- Group 3 (Active Comparator): Stainless steel crown (3M-ESPE, St. Paul, Minnesota, USA)
  Interventions: Other: Dental Crown
- Group 4 (Active Comparator): Strip Crown (3M-ESPE, St. Paul, Minnesota, USA)
  Interventions: Other: Dental Crown

INTERVENTIONS:
Other: Dental Crown — Pediatric size dental crown; restore damaged tooth to its normal shape, size, and function.
  Other Names: Zirconia Crown (NuSmile, Houston, Texas, USA); Stainless Steel Crown (3M-ESPE, St. Paul, Minnesota, USA); Strip Crown (3M-ESPE, St. Paul, Minnesota, USA)

SUMMARY:
Objective: Early loss of primary teeth due to caries, can cause occlusion disorders, aesthetic problems, nutritional problems, abnormal language habits, speech disorders and psychological problems temporary or permanent. The purpose of this study was to evaluate the success of using prefabricated aesthetic crowns for the restoration of excessive tooth loss.

Study design: In this randomized, non-blinded clinical study a total of 45 teeth were included, primary molars and anterior teeth and requiring restoration after root canal treatment. Stainless steel(SCC), zirconia(ZC) and strip(S) crowns compared clinically, radiographically and periodontally during follow up period for 6 months. Parents were asked to fill out questionnaire at the 1st and 6th months to evaluate the satisfaction level. In addition, patients' pain and discomfort level was assessed using the visual analogue scale (VAS) scale.

DETAILED DESCRIPTION:
The color of crowns made it impossible to blind during clinical assessment. Thus, this study was a non-blinded, randomised, and prospective clinical trial.

Sample size: This study included 20 maxillary anterior and 25 posterior teeth that required restoration due to excessive material loss. The study groups were:

Zirconia crown(ZC) restoration on the primary central and lateral tooth with root canal treatment (n = 10), strip crown(S) restoration on the primary central and lateral tooth with root canal treatment (n = 10), Zirconia crown(ZC) restoration on primary teeth with root canal treatment (n = 12), Stainless-steel crown(SSC) restoration on primary teeth with root canal treatment (n = 13).

Clinical Procedure:

Assessment

Clinical assesment: Table 1 Gingival scores: Löe and Silness Gingival Index(GI)[Löe, 1967].

Periapical radiographic evaluation: Preoperative and every follow up visit. (Radiographic assesment: Table 2)

Intraoral photos (standard method): before treatment, after treatment and at every follow-up visit.

Crown restoration: All caries were removed after administration of local anaesthesia and proper isolation. Calcium hydroxide/iodoform paste (Vitapex®) pulpectomy was performed according to the guideline. Teeth were restored with a composite resin Nova Resin (IMICRYL®, Konya, Turkey) and glass ionomer cement (MERON®, Voco, Germany) was used as a base material. Strip Crown Forms (3M-ESPE, St. Paul,Minnesota, USA) were used to restore teeth group SC. ZC group (NuSmile, Houston, Tex. the USA) and SCC(3M ESPE, Minnesota, USA) used.

Visual analogue scale(VAS): 0-2: no pain/discomfort 4-6:moderate 8-10: high pain/discomfort.

The child was asked to choose his/her feelings about the tooth after the procedure and in follow-up appointments. Parents were asked to complete their satisfaction surveys, including the post-op and 6-month controls for patient satisfaction assessment.

Statistical Method:

IBM® SPSS® Statistics V23 analysed data. The Mann-Whitney U and Chi-square tests were used for intergroup comparisons within the anterior and posterior regions. The Friedman and Cochrane Q tests were used for intra-group time-wise comparisons. Analysis results were presented as the median (q1-q3) and frequency (percentage). P<0.05 was considered statistically significant.

Table 1: Clinical assesment

Crown retention 0= yes 1= no

Individual modified gingival index 0= healthy 1= mild gingival bleeding with a papillus 2= severe inflammation

Plaque index 0= no plaque

1. = presence of plaque as a film in the gingival margin
2. = presence of moderate plaque
3. = plaque covering a large number of surfaces

Color change 0 = no coloring

1. = minor coloration
2. = noticeable coloration

Buccal strip crown surface 0 = no loss 1 = less than 50% loss 2 = more than 50% loss 4 = loss of the entire surface

Surface abrasion of the antagonist teeth 0= no abrasion

1. abrasion started on the incisal surface of the casps
2. abrasion more than on the casps

Position of the crowns regarding gingival margin 0= subgingival

1= supragingival

Occlusion 0= contact (marked or superficial) 1= no contact

Condition of the antagonistic tooth 0= natural tooth

1. restored tooth
2. stainless steel crown
3. aesthetic crowns

Location on the arch curve 0= normal alignment

1. with rotation
2. wrong position

Proximal contacts 0= good (floss passing)

1= weak, no contact

Table 2. Postoperative Radiographic Evaluation Criteria and Scores Radiographic evaluation of crown margins 0=good adaptation, continuity in crown contractions

1. small radiolucent area under the restoration
2. huge openings
3. loss of restoration

Radiographic evaluation 0= healthy, no pathology

1. presence of a pathology that does not require immediate treatment
2. presence of pathology requiring immediate treatment

Radiographic evaluation of pulpal treatment 0=appropriate root treatment

1. short or overflowed root treatment
2. failed pulpal treatment
3. tooth with no pulpal treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients without systemic disease The American Society of Anesthesiologists (ASA)1-2,
2. Patients under 10 years old to perform endodontic treatment for adequate root support
3. Clinical and radiographically confirmed dental caries scored international caries detection and assessment system(icdas) criteria 4-5.
4. Patient/parent approve

Exclusion Criteria:

1. Patients with systemic and mental diseases
2. Acute abscess or mobility
3. Internal or external resorption
4. Inadequate oral hygiene after oral health motivation that contraindicate root canal treatment
5. Need for endocarditis prophylaxis
6. Temporomandibular joint(TMJ) disorders, bruxism
7. Absence of antagonistic teeth

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Visual examination | 6 months follow up period
  The incidence of crown retention, gingival index, marginal crown localisation
Radiographic evaluation | 6 months follow up period
  Periapical film: the rate of radiolucency. According to the index, each tooth was categorized as having a normal periapical structure (score 1), small changes in bone structure (score 2), changes in bone structure with some mineral loss (score 3), periodontitis with well-defined radiolucent areas (score 4), or severe apical periodontitis with exacerbating features (score 5)

SECONDARY OUTCOMES:
Questionaire | 6 months follow up period
  A Visual Analogue Scale (VAS): no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) that underlie results

REFERENCES:
- [Background] Walia T, Brigi C, KhirAllah ARMM. Comparative evaluation of surface roughness of posterior primary zirconia crowns. Eur Arch Paediatr Dent. 2019 Feb;20(1):33-40. doi: 10.1007/s40368-018-0382-4. Epub 2018 Oct 20. PMID 30343392
- [Background] Seminario AL, Garcia M, Spiekerman C, Rajanbabu P, Donly KJ, Harbert P. Survival of Zirconia Crowns in Primary Maxillary Incisors at 12-, 24- and 36-Month Follow-Up. Pediatr Dent. 2019 Sep 15;41(5):385-390. PMID 31648670
- [Background] El Makawi Y, Khattab N. In Vitro Comparative Analysis of Fracture Resistance of Lithium Disilicate Endocrown and Prefabricated Zirconium Crown in Pulpotomized Primary Molars. Open Access Maced J Med Sci. 2019 Dec 13;7(23):4094-4100. doi: 10.3889/oamjms.2019.864. eCollection 2019 Dec 15. PMID 32165959
- [Background] Sonbol HN, Al-Bitar ZB, Shraideh AZ, Al-Omiri MK. Parental-caregiver perception of child oral-health related quality of life following zirconia crown placement and non-restoration of carious primary anterior teeth. Eur J Paediatr Dent. 2018 Mar;19(1):21-28. doi: 10.23804/ejpd.2018.19.01.04. PMID 29569449
- [Background] Lee JH. Guided tooth preparation for a pediatric zirconia crown. J Am Dent Assoc. 2018 Mar;149(3):202-208.e2. doi: 10.1016/j.adaj.2017.08.048. Epub 2018 Feb 1. PMID 29395008